CLINICAL TRIAL: NCT01446913
Title: Sleep Apnea in TIA/Stroke: Reducing Cardiovascular Risk With Positive Airway Pressure
Acronym: SleepTight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Indiana University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1101007811; U34HL105285-01 (NIH)
Record Dates: First submitted 2011-10-03; First posted 2011-10-05 (Estimated); Results first posted 2020-11-18 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-10

CONDITIONS: Transient Ischemic Attack; Stroke
Keywords: Sleep Apnea; CPAP adherence; behavioral adherence; stroke
MeSH Terms: conditions — Ischemic Attack, Transient; Stroke; Sleep Apnea Syndromes

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Standard Intervention group (Active Comparator): This group gets unattended sleep study, auto titrating CPAP, and standard CPAP support.
  Interventions: Device: Standard CPAP Intervention
- Enhanced CPAP intervention (Active Comparator): This group gets an unattended sleep study, autotitrating CPAP, and enhanced CPAP support.
  Interventions: Behavioral: Enhanced CPAP Intervention
- Usual Care (No Intervention): This group usual care after TIA/stroke and a sleep study at the end of the study.

INTERVENTIONS:
Device: Standard CPAP Intervention
  Arms: Standard Intervention group
Behavioral: Enhanced CPAP Intervention
  Arms: Enhanced CPAP intervention

SUMMARY:
The goal of this study is to develop a novel study design to safely and ethically conduct a long-term randomized controlled trial among patients at high risk for both sleep apnea and cardiovascular events that will examine whether effective positive airway pressure(PAP) therapy reduces cardiovascular risk. Patients with transient ischemic attack(TIA) or stroke have a high prevalence of sleep apnea(60-80%), and they are at high risk of cardiovascular events(myocardial infarction, congestive heart failure, recurrent stroke, and cardiovascular death)in the first year post event, despite current prevent strategies. Therefore, the treatment of sleep apnea may represent a novel therapeutic target to reduce cardiovascular outcomes in this high risk population.

DETAILED DESCRIPTION:
The proposed study is a randomized controlled trial among patients with transient ischemic attack (TIA) and minor stroke, comparing strategies for the diagnosis and treatment of sleep apnea with usual care over 6-12 months at 2 sites (Yale University School of Medicine and Indiana University School of Medicine). Patients with TIA and minor stroke will be randomly assigned to either usual care or a diagnosis and treatment approach that includes ambulatory polysomnography and initiation of autotitrating CPAP for sleep apnea in a 1:2 (control:intervention) randomization scheme. Intervention patients with sleep apnea will receive either a standard CPAP treatment intervention or an enhanced protocol designed to increase long-term CPAP adherence. The primary outcomes will include: (a) the impact of CPAP on pathophysiologic markers in the following domains of cardiovascular risk: inflammation (CRP, Il-6), heightened sympathetic activity/parasympathetic withdrawal (plasma catecholamines and heart rate variability (HRV)), insulin resistance (HOMA-IR, HbA1C), endothelial injury (flow mediated vasodilation), and atherosclerosis (carotid intima-media thickness); and (b) long-term (6-12 month) CPAP adherence.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* TIA or ischemic stroke
* within 1 week of neurological symptom onset
* brain imaging within 24 hours

Exclusion Criteria:

* known to have sleep apnea
* suspected sleep disorder other than sleep apnea
* hospice patients or patients receiving comfort only measures
* patients unable to use a nasal or face mask
* patients who require mechanical ventilation
* Non English language patients
* inability to provide informed consent
* active suicidal ideation
* live outside the recruitment area
* provider does not allow researcher to contact patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2011-05; Primary Completion 2013-12 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry Yaggi, MD,MPH, Principal Investigator — Yale University; Dawn M Bravata, M.D., Principal Investigator — Indiana University School of Medicine
Locations (2):
- United States (2):
  - Yale University, New Haven, Connecticut
  - University of Indiana, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: Yes
Resource sharing plan In compliance NIH recommendations, we affirm our commitment to share our final research data in a timely fashion for this proposed study with the scientific community. We intend this to occur no later than the time of acceptance for publication of the main findings from the final dataset. We will share all data from the funded research that can be shared without compromising individual subjects' rights and privacy, regardless of whether the data have been used for publication.

REFERENCES:
- [Background] Koo BB, Bravata DM, Tobias LA, Mackey JS, Miech EJ, Matthias MS, Stahl SM, Sico JJ, Vaz Fragoso CA, Williams LS, Lampert R, Qin L, Yaggi HK. Observational Study of Obstructive Sleep Apnea in Wake-Up Stroke: The SLEEP TIGHT Study. Cerebrovasc Dis. 2016;41(5-6):233-41. doi: 10.1159/000440736. Epub 2016 Jan 27. PMID 26811929
- [Derived] Yaggi HK, Mittleman MA, Bravata DM, Concato J, Ware J, Stoney CM, Redline S. Reducing cardiovascular risk through treatment of obstructive sleep apnea: 2 methodological approaches. Am Heart J. 2016 Feb;172:135-43. doi: 10.1016/j.ahj.2015.07.033. Epub 2015 Sep 11. PMID 26856225

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three patients withdrew prior to randomization.
Groups:
- Standard Intervention Group: This group gets unattended sleep study, auto titrating CPAP, and standard CPAP support.
  Standard CPAP Intervention
- Enhanced CPAP Intervention: This group gets an unattended sleep study, autotitrating CPAP, and enhanced CPAP support.
  Enhanced CPAP Intervention
Period: Overall Study
Arm/Group | Standard Intervention Group | Enhanced CPAP Intervention | Usual Care
Started | 86 | 82 | 84
Patients With Sleep Study (A sub sample of patients had a valid sleep study conducted.) | 53 | 56 | 29
Patients With Sleep Apnea (A sub sample of patients with sleep apnea were studied.) | 39 | 45 | 21
Completed | 77 | 73 | 73
Not Completed | 9 | 9 | 11
Not completed — Significant illness | 1 | 1 | 1
Not completed — Withdrawal by Subject | 5 | 3 | 5
Not completed — Physician Decision | 0 | 0 | 2
Not completed — Lost to Follow-up | 3 | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Intervention Group | Enhanced CPAP Intervention | Usual Care | Total
Number analyzed (Participants) | 86 | 82 | 84 | 252
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 60 | 59 | 61 | 180
  >=65 years | 26 | 23 | 23 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (12.5) | 61.3 (12.8) | 60.3 (12.5) | 60.5 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 37 | 42 | 121
  Male | 44 | 45 | 42 | 131
Region of Enrollment [Number; unit: participants]
  United States | 86 | 82 | 84 | 252

OUTCOME MEASURES:

1. Primary Outcome: HOMA IR Change From Baseline
Description: The homeostasis model assessment-estimated insulin resistance (HOMA-IR). HOMA IR change is one of the measures used to assess cardiovascular risk. HOMA-IR Index (measured by calculating - fasting insulin (microU/L) x fasting glucose (nmol/L)/22.5.). The change from baseline up until the final measurement (up to 12 months) was assessed.
Time Frame: Baseline and up to 12 months
Population: Intention to treat analysis population.
Measure: Mean (Standard Deviation); unit: HOMA-IR Index
Arm/Group | Standard Intervention Group | Enhanced CPAP Intervention | Usual Care
Number analyzed (Participants) | 86 | 82 | 84
HOMA-IR Index | 0.9 (3.0) | 4.0 (12.7) | 4.1 (24.8)

2. Primary Outcome: CRP Change From Baseline
Description: C-reactive protein (CRP) is a blood test marker for inflammation in the body. CRP is produced in the liver and its level is measured by testing the blood. CRP is classified as an acute phase reactant, which means that its levels will rise in response to inflammation. CRP is one of the measures used to assess cardiovascular risk. The change from baseline up until the final measurement (up to 12 months) was assessed.
Time Frame: Baseline and up to 12 months
Population: Intention to treat analysis.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Standard Intervention Group | Enhanced CPAP Intervention | Usual Care
Number analyzed (Participants) | 86 | 82 | 84
mg/dl | 0.8 (14.4) | 0.9 (10.2) | -3.0 (13.0)

3. Primary Outcome: IL-6 Change From Baseline
Description: IL-6 is a type of protein known as a cytokine, produced by cells of the immune system in response to an infection. IL-6 test results measure the amount of IL-6 circulating in the blood and are used as one sign of systemic inflammation. Il-6 is one of the measures used to assess cardiovascular risk. The change from baseline up until the final measurement (up to 12 months) was assessed.
Time Frame: Baseline and up to 12 months
Population: Intention to treat analysis.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Standard Intervention Group | Enhanced CPAP Intervention | Usual Care
Number analyzed (Participants) | 86 | 82 | 84
pg/ml | 4.0 (11) | 1.8 (40.6) | -0.7 (3.9)

4. Primary Outcome: Catecholamine Change From Baseline
Description: Catecholamine testing measures the amounts of catecholamines which are a group of similar substances/hormones released into the blood in response to physical or emotional stress. The primary catecholamines are dopamine, epinephrine (adrenaline), and norepinephrine. Catecholamine is one of the measures used to assess cardiovascular risk. The change from baseline up until the final measurement (up to 12 months) was assessed.
Time Frame: Baseline and up to 12 months
Population: Intention to treat analysis.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Standard Intervention Group | Enhanced CPAP Intervention | Usual Care
Number analyzed (Participants) | 86 | 82 | 84
pg/ml | 192.4 (385.0) | 5.8 (259.6) | 89.0 (231.8)

5. Primary Outcome: Heart Rate Variability Change From Baseline
Description: Heart rate variability (HRV) is the constant variation in milliseconds between heartbeats. HRV is one of the measures used to assess cardiovascular risk. The change from baseline up until the final measurement (up to 12 months) was assessed.
Time Frame: Baseline and up to 12 months
Population: Intention to treat analysis.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Standard Intervention Group | Enhanced CPAP Intervention | Usual Care
Number analyzed (Participants) | 86 | 82 | 84
milliseconds | -8.0 (20.0) | 5.0 (30.5) | -1.5 (26.4)

6. Primary Outcome: 24-H Systolic Blood Pressure Mean Change From Baseline
Description: 24-H Systolic Blood Pressure is one of the measures used to assess cardiovascular risk- this was assessed multiple times and averaged across a in 24 hour time period. The change from baseline up until the final measurement (up to 12 months) was assessed.
Time Frame: Baseline and up to 12 months
Population: Intention to treat analysis.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Standard Intervention Group | Enhanced CPAP Intervention | Usual Care
Number analyzed (Participants) | 86 | 82 | 84
mmHg | 0.6 (12.8) | -1.2 (12.5) | 5.9 (13.4)

7. Primary Outcome: Flow-mediated Vasodilation Mean Change From Baseline
Description: Flow-mediated vasodilation is performed when the brachial artery diameter is measured (in mm) during three conditions; baseline (after at least 10 min supine rest), during reactive hyperaemia (induced by inflation to 250 mmHg and then deflation of a sphygmomanometer cuff around the forearm) and finally after the administration of sublingual nitroglycerin. A linear array, high resolution ultrasound transducer is used to provide B-mode images of the target vessel, proximal to the forearm cuff. Flow-mediated vasodilation is one of the measures used to assess cardiovascular risk and the mean of the change in the multiple measurements was used at each time point. The change from baseline up until the final measurement (up to 12 months) was assessed.
Time Frame: Baseline to up to 12 months
Population: Intention to treat analysis.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Standard Intervention Group | Enhanced CPAP Intervention | Usual Care
Number analyzed (Participants) | 86 | 82 | 84
mm | 1.0 (3.0) | 0.1 (2.2) | -0.3 (2.9)

8. Primary Outcome: Carotid Intima-Medial Thickness Mean Change From Baseline
Description: Carotid Intima-Medial Thickness are measurements of the mean values of Intima-media thickness (IMT) of carotid arteries. Caroid Intima-Medial Thickness mean change is one of the measures used to assess cardiovascular risk. The change from baseline up until the final measurement (up to 12 months) was assessed.
Time Frame: Baseline to up to 12 months
Population: Intention to treat analysis.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Standard Intervention Group | Enhanced CPAP Intervention | Usual Care
Number analyzed (Participants) | 86 | 82 | 84
mm | 0.0 (0.1) | 0.0 (0.1) | 0.0 (0.1)

9. Primary Outcome: CPAP Adherence Rates Change From Baseline
Description: CPAP adherence rates were calculated as hours of CPAP use per night. The change from baseline up until the final measurement (up to 12 months) was assessed. The Respironics M-series (now System One, Phillips Respironics, North Ryde, Australia) produced a record of the patient adherence (hours of use per night) throughout the duration of the follow up period.
Time Frame: Baseline to up to 12 months
Population: The analysis population is a subset of patients in the standard and enhanced intervention arms that had a diagnosis of sleep apnea.
Measure: Mean (Standard Deviation); unit: Hours per night
Groups:
- Standard: Standard Intervention patients with a diagnosis of sleep apnea.
- Enhanced: Enhanced Intervention patients with a diagnosis of sleep apnea.
Arm/Group | Standard | Enhanced
Number analyzed (Participants) | 39 | 45
Hours per night | 3.9 (2.1) | 4.3 (2.4)

10. Secondary Outcome: HOMA IR Change From Baseline With CPAP Use
Description: The homeostasis model assessment-estimated insulin resistance (HOMA-IR). HOMA IR change is one of the measures used to assess cardiovascular risk. HOMA-IR Index (measured by calculating - fasting insulin (microU/L) x fasting glucose (nmol/L)/22.5.) To determine if CPAP use had an impact on cardiovascular risk, these measures were compared among CPAP usage groups. The change from baseline up until the final measurement (up to 12 months) was assessed.
Time Frame: Baseline to up to 12 months
Population: The analysis population comprises of those with a sleep apnea diagnosis from a valid sleep study and is split into 3 categories of CPAP use where the treatment arms are combined.
Measure: Mean (Standard Deviation); unit: HOMA-IR Index
Groups:
- No CPAP Use: Intervention and control patients with none/poor CPAP use
- Some CPAP Use: Intervention patients with some CPAP (less than 4 hours per night)
- Good CPAP Use: Intervention patients with good CPAP use (>=4 hours per night)
Arm/Group | No CPAP Use | Some CPAP Use | Good CPAP Use
Number analyzed (Participants) | 39 | 26 | 32
HOMA-IR Index | -0.2 (1.0) | 2.4 (12.0) | 3.3 (9.7)

11. Secondary Outcome: CRP Change From Baseline With CPAP Use
Description: C-reactive protein (CRP) is a blood test marker for inflammation in the body. CRP is produced in the liver and its level is measured by testing the blood. CRP is classified as an acute phase reactant, which means that its levels will rise in response to inflammation. CRP is one of the measures used to assess cardiovascular risk. To determine if CPAP use had an impact on cardiovascular risk, these measures were compared among CPAP usage groups. The change from baseline up until the final measurement (up to 12 months) was assessed.
Time Frame: Baseline to up to 12 months
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | No CPAP Use | Some CPAP Use | Good CPAP Use
Number analyzed (Participants) | 39 | 26 | 32
mg/dl | 0.8 (14.4) | 0.9 (10.2) | -3.0 (13.0)

12. Secondary Outcome: IL-6 Change From Baseline With CPAP Use
Description: IL-6 is a type of protein known as a cytokine, produced by cells of the immune system in response to an infection. IL-6 test results measure the amount of IL-6 circulating in the blood and are used as one sign of systemic inflammation. IL-6 is one of the measures used to assess cardiovascular risk. To determine if CPAP use had an impact on cardiovascular risk, these measures were compared among CPAP usage groups. The change from baseline up until the final measurement (up to 12 months) was assessed.
Time Frame: Baseline to up to 12 months
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | No CPAP Use | Some CPAP Use | Good CPAP Use
Number analyzed (Participants) | 39 | 26 | 32
pg/ml | -5.3 (27.3) | 3.3 (11.5) | 11.9 (41.7)

13. Secondary Outcome: Catecholamine Change From Baseline With CPAP Use
Description: Catecholamine testing measures the amounts of catecholamines which are a group of similar substances/hormones released into the blood in response to physical or emotional stress. The primary catecholamines are dopamine, epinephrine (adrenaline), and norepinephrine. Catecholamines change is one of the measures used to assess cardiovascular risk. To determine if CPAP use had an impact on cardiovascular risk, these measures were compared among CPAP usage groups. The change from baseline up until the final measurement (up to 12 months) was assessed.
Time Frame: Baseline to up to 12 months
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | No CPAP Use | Some CPAP Use | Good CPAP Use
Number analyzed (Participants) | 39 | 26 | 32
pg/ml | 76.7 (245.5) | -27.8 (288.2) | 184 (436.6)

14. Secondary Outcome: Heart Rate Variability Change From Baseline With CPAP Use
Description: Heart rate variability (HRV) is the constant variation in milliseconds between heartbeats. HRV is one of the measures used to assess cardiovascular risk. To determine if CPAP use had an impact on cardiovascular risk, these measures were compared among CPAP usage groups. The change from baseline up until the final measurement (up to 12 months) was assessed.
Time Frame: Baseline to up to 12 months
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | No CPAP Use | Some CPAP Use | Good CPAP Use
Number analyzed (Participants) | 39 | 26 | 32
milliseconds | 3.2 (18.9) | -5.4 (24.8) | 5.3 (33.5)

15. Secondary Outcome: 24-H Mean Systolic Blood Pressure Change From Baseline With CPAP Use
Description: 24-H Mean Systolic Blood Pressure change is one of the measures used to assess cardiovascular risk- this was assessed multiple times and averaged across a in 24 hour time period. To determine if CPAP use had an impact on cardiovascular risk, these measures were compared among CPAP usage groups. The change from baseline up until the final measurement (up to 12 months) was assessed.
Time Frame: Baseline to up to 12 months
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | No CPAP Use | Some CPAP Use | Good CPAP Use
Number analyzed (Participants) | 39 | 26 | 32
mmHg | 3.8 (11.1) | -4.9 (15.0) | 0.1 (10.3)

16. Secondary Outcome: Flow-mediated Vasodilation Mean Change From Baseline With CPAP Use
Description: Flow-mediated vasodilation is performed when the brachial artery diameter is measured (in mm) during three conditions; baseline (after at least 10 min supine rest), during reactive hyperaemia (induced by inflation to 250 mmHg and then deflation of a sphygmomanometer cuff around the forearm) and finally after the administration of sublingual nitroglycerin. A linear array, high resolution ultrasound transducer is used to provide B-mode images of the target vessel, proximal to the forearm cuff. Flow-mediated vasodilation is one of the measures used to assess cardiovascular risk and the mean of the change in the multiple measurements was used at each time point. To determine if CPAP use had an impact on cardiovascular risk, these measures were compared among CPAP usage groups. The change from baseline up until the final measurement (up to 12 months) was assessed.
Time Frame: Baseline to up to 12 months
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | No CPAP Use | Some CPAP Use | Good CPAP Use
Number analyzed (Participants) | 39 | 26 | 32
mm | -0.7 (3.2) | 2.7 (3.1) | 0.3 (2.1)

17. Secondary Outcome: Carotid Intima-Medial Thickness Change From Baseline With CPAP Use Change
Description: Carotid Intima-Medial Thickness are measurements of the mean values of Intima-media thickness (IMT) of carotid arteries. Caroid Intima-Medial Thickness change is one of the measures used to assess cardiovascular risk. To determine if CPAP use had an impact on cardiovascular risk, these measures were compared among CPAP usage groups. The change from baseline up until the final measurement (up to 12 months) was assessed. The carotid intimal thickness measurement was obtained by averaging the distance between the lumen-intima interface and the media-adventitia interface obtained from 5 contiguous sites 1 mm apart.
Time Frame: Baseline to up to 12 months
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | No CPAP Use | Some CPAP Use | Good CPAP Use
Number analyzed (Participants) | 39 | 26 | 32
mm | 0.0 (0.1) | 0.0 (0.1) | 0.0 (0.1)

18. Secondary Outcome: Medication-adjusted 24-H SBP Change From Baseline
Description: Change in medication-adjusted 24-hour SBP, which is calculated as [mean 24-hour SBP in mmHg] + [patient's DDD × (8.0 mmHg), was assessed between CPAP adherence groups. The change from baseline up until the final measurement (up to 12 months) was assessed.
Time Frame: Baseline to up to 12 months
Population: The analysis population comprises of those with a sleep apnea diagnosis and is split into 3 categories of CPAP use where the treatment arms are combined.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | No CPAP Use | Some CPAP Use | Good CPAP Use
Number analyzed (Participants) | 39 | 26 | 32
mmHg | 7.8 (13.9) | 5.3 (17.3) | 0.1 (12.3)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored through the 12 month follow up period.
Arm/Group | Standard Intervention Group | Enhanced CPAP Intervention | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/86 | 4/82 | 2/84
Serious Adverse Events (participants affected / at risk) | 3/86 | 6/82 | 7/84
Other Adverse Events (participants affected / at risk) | 2/86 | 3/82 | 3/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Intervention Group (N=86) | Enhanced CPAP Intervention (N=82) | Usual Care (N=84)
Recurrent Stroke (Nervous system disorders) | 1 (1) | 5 (6) | 6 (6) — Recurrent stroke
acute MI (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — acute MI
Unstable angina hospitalization (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) — Unstable angina hospitalization
Urgent coronary revascularization (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) — coronary revascularization
Stroke (Nervous system disorders) | 1 (1) | 5 (5) | 6 (6)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Intervention Group (N=86) | Enhanced CPAP Intervention (N=82) | Usual Care (N=84)
Falls (General disorders) | 2 (2) | 3 (3) | 3 (3) — falls

LIMITATIONS AND CAVEATS:
A study design which compares the effectiveness of a diagnostic and treatment strategy to usual care may result in an underestimate of the efficacy and potency of CPAP on our outcomes. Not all patients in the intervention strategy had sleep apnea.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No